CLINICAL TRIAL: NCT03465176
Title: The Effect of Aroma on Fatigue Scores Among Women With Hypothyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1600
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Fatigue; Hypothyroidism
Keywords: aromatherapy; fatigue; hypothyroidism; essential oils
MeSH Terms: conditions — Fatigue; Hypothyroidism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The women in this arm will receive an essential oil blend to inhale each afternoon for two weeks.
  Interventions: Other: Aromatherapy Blend
- Control (Placebo Comparator): The women in this arm will receive an odorless vegetable based oil to inhale each afternoon for two weeks as a control/placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Aromatherapy Blend — The essential oil intervention is a blend of plant derived oils which have been distilled from crude plant matter and analyzed in a laboratory to identify chemical composition.
  Arms: Intervention
Other: Placebo — The placebo substance is an odorless vegetable oil derived from avocados.
  Arms: Control

SUMMARY:
This study evaluates the effects of an inhaled blend of essential oils on fatigue scores among women who have hypothyroidism. Half of the participants will receive an essential oil blend to inhale daily for two weeks while the other half will serve as controls and inhale a carrier oil.

DETAILED DESCRIPTION:
The inhalation of certain essential oils has been found to increase stamina and reduce fatigue among athletes but have not been evaluated for the purpose of reducing fatigue among women who experience fatigue as a result of a hypothyroid condition.

The essential oils used in this study are inhaled mid-afternoon, the time in which women with hypothyroidism typically experience the lowest levels of energy during the day, otherwise known as the "afternoon slump." The essential oil is administered during this time to evaluate both the immediate effects on fatigue as well as the overall effects, with measurements at the end of both the first and second week of the study.

Fatigue is measured on a multi-dimensional scale, a validated instrument that measures not only physical fatigue but also emotional and mental fatigue.

ELIGIBILITY:
Inclusion Criteria:

* female
* diagnosed with hypothyroidism
* otherwise healthy

Exclusion Criteria:

• history of thyroid cancer

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
83-item Multidimensional Symptoms of Fatigue Inventory | 2 weeks
  This measurement collects self reported fatigue scores at baseline and at the end of each week of the intervention. Each item is scored from 0-4, with higher scores indicating greater levels of fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Franklin Institute of Wellness, Franklin, Tennessee, United States